CLINICAL TRIAL: NCT01995136
Title: Investigation of the Effect of Travoprost Ophthalmic Solution of Lowering Intraocular Pressure in Patients With Normal Tension Glaucoma
Brief Title: Investigation of Intraocular Pressure (IOP) Reduction Efficacy of Travoprost Ophthalmic Solution in Patients With Normal Tension Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-13-047; UMIN000011621 (Registry Identifier: UMIN)
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Normal Tension Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular hypertension
MeSH Terms: conditions — Low Tension Glaucoma; Ocular Hypertension; Glaucoma | interventions — Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRAVATAN Z (Experimental): Travoprost Ophthalmic Solution 0.004%, 1 drop instilled in each eye once daily at 9PM for 3 months.
  Interventions: Drug: Travoprost Ophthalmic Solution 0.004%

INTERVENTIONS:
Drug: Travoprost Ophthalmic Solution 0.004% — benzalkonium chloride (BAC) free
  Other Names: TRAVATAN Z®

SUMMARY:
The purpose of this study is to investigate IOP reduction efficacy of travoprost 0.004% ophthalmic solution (TRAVATAN Z®) in subjects with normal tension glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of normal tension glaucoma.
* Must sign an Informed Consent form.
* IOP within protocol-specified range.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Pregnant and lactating women, or women who intend to become pregnant during the study period.
* Advanced and serious glaucoma, as specified in protocol.
* Complicated chronic or recurrent uveitis, scleritis or corneal herpes.
* History of ocular trauma, intraocular surgery or laser surgery for the included eye.
* Ocular-infection and severe ocular complication.
* Best-corrected visual acuity (BCVA) worse than 0.2 decimal.
* Difficulty in conducting applanation tonometry for the included eye as determined by the doctor.
* Severe or serious hypersensitivity to prostaglandin analogues or any ingredients used in the study.
* Use of IOP lowering ophthalmic solutions other than TRAVATAN Z® or oral carbonic anhydrase inhibitor (Diamox, etc.) during the study period.
* Use of any adrenocorticosteroids during the study period.
* Use of IOP lowering ophthalmic solution within the past 30 days.
* Regarded by doctor as not suitable for study participation.
* Other protocol-specified exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danyel Carr, MS, Study Director — Alcon Japan, Ltd.
Locations (1):
- Alcon Japan, Ltd., Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 study sites located in Japan.
Pre-assignment Details: This reporting group includes all enrolled subjects (32).
Groups:
- TRAVATAN Z: Ophthalmic Solution, 1 drop instilled in each eye once daily at 9PM for 3 months.
Period: Overall Study
Arm/Group | TRAVATAN Z
Started | 32
Completed | 31
Not Completed | 1
Not completed — Change in residence | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled subjects minus any subjects with all missing data and/or critical protocol deviation/s.
Arm/Group | TRAVATAN Z
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Baseline IOP [Mean (Standard Deviation); unit: mmHg]
  9:00 AM | 16.55 (1.43)
  1:00 PM | 15.72 (1.82)
  5:00 PM | 15.73 (2.17)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in IOP (9:00 AM) at Week 4, Week 8, and Week 12
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in millimeters of mercury (mmHg). Data at 9:00 AM from Weeks 4, 8, and 12 were pooled. A more negative change indicates a greater amount of improvement. One eye (study eye) was subject to analysis.
Time Frame: Baseline (Day 0), Week 4, Week 8, Week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | TRAVATAN Z
Number analyzed (Participants) | 30
mmHg
  Baseline | 16.55 [15.88 to 17.22]
  Change from Baseline | -3.37 [-3.90 to -2.85]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (Sep 2013 - Jun 2014). This analysis population includes all subjects enrolled in the study, minus any subject whose safety evaluation data is all missed (1 subject).
Description: An AE was defined as any medically undesirable event that develops in a subject that received the study drug regardless of causal relationship with the study drug.
Arm/Group | TRAVATAN Z
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.